CLINICAL TRIAL: NCT06580912
Title: Krill Oil for Pain and Physical Function in Older Adults
Brief Title: Krill Oil for Pain in Elders
Acronym: KOPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB202400581; P30AG028740 (NIH)
Record Dates: First submitted 2024-08-26; First posted 2024-08-30 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-02

CONDITIONS: Chronic Musculoskeletal Pain
Keywords: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Krill oil (Experimental): 4 grams of krill oil per day
  Interventions: Drug: Krill oil
- Mixed vegetable oil (Placebo Comparator): 4 grams of mixed vegetable oil per day
  Interventions: Dietary Supplement: Mixed vegetable oil

INTERVENTIONS:
Drug: Krill oil — 4 grams of krill oil per day
  Arms: Krill oil
Dietary Supplement: Mixed vegetable oil — 4 grams of mixed vegetable oil per day
  Arms: Mixed vegetable oil

SUMMARY:
Chronic musculoskeletal pain contributes to mobility disability among older adults. Nutritional interventions, like omega-3 fatty acids, may help manage pain and improve physical function. Supplementation with krill oil may offer advantages to fish oil due to better absorption and additional nutrients. This pilot study aims to assess the feasibility of a clinical trial to determine the impact of krill oil supplementation on pain and function in older adults, informing future research.

DETAILED DESCRIPTION:
Mobility is a critical factor in the maintenance of independence and quality of life of older adults. Chronic musculoskeletal pain contributes to mobility disability disproportionately among older adults. Current treatments for pain and functional decline are often ineffective and add to heightened risks of polypharmacy in older adults. As such, nutritional interventions can play a significant role in promoting health and longevity, managing pain, and enhancing physical function in older adults. Omega (ω)-3 polyunsaturated fatty acids (PUFAs) are essential nutrients that are well recognized for their anti-inflammatory and cardioprotective benefits, as well as their analgesic and anti-nociceptive properties. Most American adults do not meet the recommendations for ω-3 intakes, particularly eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), found primarily in seafood. Due to competing pathways, an elevated ω-6 to ω-3 ratio contributes to an overproduction of pro-inflammatory eicosanoids and the development of chronic diseases. A high ω-6:ω-3 ratio is associated with higher chronic pain prevalence and increased pain severity. Additionally, ω-3 PUFAs may play a role in the preservation of muscle and physical function in older adults. Low levels of ω-3s in blood are associated with reduced muscle strength, slower gait speed, and mobility disability among older adults. Considered largely safe and cost-effective, ω-3 supplementation may be crucial to increasing the intake of these essential nutrients and achieving optimal levels among older adults. Although the use of EPA and DHA has been incorporated into several guidelines, a scarcity of data has prevented the development of strong recommendations on the use of ω-3 supplementation for the maintenance of physical function in older adults, particularly those with chronic musculoskeletal pain. Krill oil has been recently proposed as an advantageous alternative to traditional fish oil supplements, due to a greater bioavailability of EPA and DHA and additional bioactive compounds. The goal of the proposed pilot study is to assess the feasibility of a 3-month randomized controlled trial to determine the effectiveness of krill oil supplementation on pain and physical function in older adults with chronic musculoskeletal pain. The investigators will enroll 40 older adults (≥60 years) who will be randomly assigned to 4 g krill oil (1,288 mg/d EPA+DHA, 0.45 mg astaxanthin, 320 mg choline) daily or matched placebo (mixed lipids without EPA and DHA). The investigators will determine the impact of krill oil supplementation on the omega-3 index (%EPA+DHA in erythrocytes), the ω-6/ω-3 ratio, and inflammatory biomarkers in blood, and obtain preliminary evidence of its impact on pain and physical function in older adults. The findings of this pilot will inform a future fully-powered randomized controlled trial by assessing the feasibility and acceptability of krill oil supplementation among older U.S. adults with chronic musculoskeletal pain.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged ≥60 years
* Exhibiting chronic musculoskeletal pain of the hip, knees, or lower back (>3 months)
* Average pain ≥4 on a 0-10 numeric rating scale
* Exhibiting moderate mobility limitations (Short Physical Performance Battery score 4-10)
* Ability to take oral supplements and be willing to adhere to the supplementation regimen
* Agreement to adhere to Lifestyle Considerations throughout study duration

Exclusion Criteria:

* Any known coagulation or bleeding disorders
* Standing regimen of anticoagulants or full-dose aspirin
* Regular use of opioids or high-dose NSAIDs
* Taking medication known to affect muscle (e.g. steroids)
* Taking selective serotonin reuptake inhibitors (SSRIs)
* Omega-3 supplementation within the past 3 months
* High consumption of fatty fish (>2 servings/week)
* Habitual supplementation with other complementary medicines/supplements that may affect the study results, including St. John's Wort
* Known allergy to seafood
* Clinically significant conditions: diabetes, severe cardiovascular disease, seizure disorders, uncontrolled hypertension (>150/90mmhg at baseline), cancer or cancer that has been in remission >5 years
* History of atrial fibrillation or atrial flutter
* Dementia
* History of smoking, alcohol abuse, or illicit drug use
* Ambulatory impairments which would limit the ability to perform physical function tests
* Treatment with another investigational drug or other intervention within 3 months
* Planning a surgical procedure during the study period
* Planning to permanently leave the area during the study period

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-17 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Omega-3 Index | Baseline, 6 weeks, and 12 weeks
  Percent EPA+DHA in erythrocytes
Graded Chronic Pain Scale-Revised (GCPS-R) | Baseline, 6 weeks, and 12 weeks
  An updated version of the original Graded Chronic Pain Scale (GCPS), a widely used tool in pain research and clinical settings. The GCPS-R assesses the severity and impact of chronic pain by measuring pain intensity and pain-related disability. The scale provides a disability score, which classifies individuals into different levels of pain-related disability. The GCPS-R is useful for both screening and monitoring chronic pain.
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Baseline, 6 weeks, and 12 weeks
  Well-validated and widely utilized measure of pain symptoms and physical disability. It is comprised of 24 items to evaluate three domains: pain, stiffness, and physical function. Responses can be summated for domain-specific scores, as well as a global score.
Short Physical Performance Battery (SPPB) | Baseline and 12 weeks
  Widely used geriatric assessment designed to evaluate the physical performance and mobility of older adults. It consists of a series of simple tests that assess three major components: balance, gait speed, and lower extremity strength (chair stand test). Each component is scored on a scale from 0 to 4, with higher scores indicating better performance. An SPPB of ≤10 is predictive of mobility disability and all-cause mortality.
6-Minute Walk Test (6MWT) | Baseline and 12 weeks
  Simple, inexpensive, sub-maximal exercise test commonly used to assess functional capacity and endurance in older adults. Participants are instructed to cover as much distance as possible in 6 minutes along a rectangular pathway. Normative data for 6MWT performance by age in older adults is available for comparison.
Handgrip Strength Test (HGST) | Baseline and 12 weeks
  Handgrip strength is a measure of physical function and is suggested as a biomarker of aging. Maximal grip strength for each hand will be measured using a handheld dynamometer.

SECONDARY OUTCOMES:
Inflammatory Biomarkers | Baseline and 12 weeks
  The investigators will evaluate concentrations of inflammatory biomarkers, including but not limited to high-sensitivity C-reactive protein, interleukin-6, and tumor necrosis factors-alpha from blood samples.
Patient Global Impression of Change (PGIC) | 6 weeks and 12 weeks
  Self-reported measure that assesses a patient's overall perception of improvement or decline in their condition following treatment. It is typically used in clinical trials to gauge the efficacy of an intervention from the patient's perspective, with responses ranging from "very much improved" to "very much worse."
Medicine Acceptability Questionnaire (MAQ) | 6 weeks and 12 weeks
  Tool designed to assess patients' perceptions and experiences of taking medications. It evaluates factors such as ease of use, taste, and overall satisfaction, providing insights into patient adherence and preferences.
Pepper Assessment Tool for Disability (PAT-D) | Baseline and 12 weeks
  23-item instrument measuring 5 domains of function in older adults: mobility, transferring, upper extremity, activities of daily living (ADL), and instrumental activities of daily living (IADL).
Montreal Cognitive Assessment (MoCA) | Screening, 6 weeks, and 12 weeks
  Brief, 10-minute measure of global cognitive function and a screening tool for mild-to-severe cognitive impairment. The test assesses cognitive domains, such as attention, memory, orientation, language, conceptual thinking, and planning. Different versions of the MoCA will be used at each visit to minimize retest effects.
NIH Toolbox Cognition Battery | Baseline and 12 weeks
  The NIH Toolbox Cognition Battery is comprised of 7 tests that measure 8 abilities within 6 major cognitive domains: executive function, episodic memory, language, processing speed, working memory, and attention. Composite scores will be calculated for (1) fluid, (2) crystallized, and (3) global cognitive function.
Fear Avoidance Beliefs Questionnaire (FABQ) | Baseline and 12 weeks
  Self-report tool used to assess the extent to which individuals with musculoskeletal pain, particularly lower back pain, avoid physical activity and work due to fear that it will exacerbate their pain. It helps identify patients who may be at risk of developing chronic pain due to fear-avoidance behaviors.
EuroQol 5 Dimension 5 Level (EQ-5D-5L) | Baseline and 12 weeks
  The EQ-5D-5L is a standardized instrument used to measure health-related quality of life. It includes five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with five levels of severity, allowing for a detailed assessment of an individual's overall health status.
Brief Pittsburgh Sleep Quality Index (B-PSQI) | Baseline and 12 weeks
  A shortened version of the original Pittsburgh Sleep Quality Index, designed to quickly assess sleep quality over a one-month period. It measures aspects like sleep duration, sleep disturbances, and daytime dysfunction.
Pain Self-Efficacy Questionnaire | Baseline and 12 weeks
  10-item tool used to assess the confidence of individuals with chronic pain in performing daily activities despite their pain. It evaluates how much they believe they can manage or cope with their pain in various situations, providing insights into their psychological resilience and ability to function.
Perceived Stress Scale (PSS) | Baseline and 12 weeks
  Psychological tool used to measure the degree to which individuals perceive situations in their lives as stressful. It assesses feelings of stress over the past month, focusing on how unpredictable, uncontrollable, and overloaded respondents find their lives.
Geriatric Depression Scale-Short Form | Baseline and 12 weeks
  15-item screening tool designed to assess depression in older adults. It is a simplified version of the original Geriatric Depression Scale and is commonly used due to its brevity and effectiveness in identifying depressive symptoms in elderly populations.

CONTACTS AND LOCATIONS:
Overall Officials: Javier A Tamargo, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Claude D. Pepper Older Americans Independence Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sibille KT, King C, Garrett TJ, Glover TL, Zhang H, Chen H, Reddy D, Goodin BR, Sotolongo A, Petrov ME, Cruz-Almeida Y, Herbert M, Bartley EJ, Edberg JC, Staud R, Redden DT, Bradley LA, Fillingim RB. Omega-6: Omega-3 PUFA Ratio, Pain, Functioning, and Distress in Adults With Knee Pain. Clin J Pain. 2018 Feb;34(2):182-189. doi: 10.1097/AJP.0000000000000517. PMID 28542024
- [Background] Stonehouse W, Benassi-Evans B, Bednarz J, Vincent AD, Hall S, Hill CL. Krill oil improved osteoarthritic knee pain in adults with mild to moderate knee osteoarthritis: a 6-month multicenter, randomized, double-blind, placebo-controlled trial. Am J Clin Nutr. 2022 Sep 2;116(3):672-685. doi: 10.1093/ajcn/nqac125. PMID 35880828
- [Background] Suzuki Y, Fukushima M, Sakuraba K, Sawaki K, Sekigawa K. Krill Oil Improves Mild Knee Joint Pain: A Randomized Control Trial. PLoS One. 2016 Oct 4;11(10):e0162769. doi: 10.1371/journal.pone.0162769. eCollection 2016. PMID 27701428
- [Background] Alkhedhairi SA, Aba Alkhayl FF, Ismail AD, Rozendaal A, German M, MacLean B, Johnston L, Miller AA, Hunter AM, Macgregor LJ, Combet E, Quinn TJ, Gray SR. The effect of krill oil supplementation on skeletal muscle function and size in older adults: A randomised controlled trial. Clin Nutr. 2022 Jun;41(6):1228-1235. doi: 10.1016/j.clnu.2022.04.007. Epub 2022 Apr 20. PMID 35504165
- [Background] Laslett LL, Scheepers LEJM, Antony B, Wluka AE, Cai G, Hill CL, March L, Keen HI, Otahal P, Cicuttini FM, Jones G. Krill Oil for Knee Osteoarthritis: A Randomized Clinical Trial. JAMA. 2024 Jun 18;331(23):1997-2006. doi: 10.1001/jama.2024.6063. PMID 38776073

DOCUMENTS (1):
  • Informed Consent Form (2025-07-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT06580912/ICF_000.pdf